CLINICAL TRIAL: NCT02170935
Title: Multicenter, Open-label-study to Assess PK Profile of a Single Oral Dose of 150 mg BIBR 1048 (Capsule) in Patients Shortly After Primary Elective Total Hip Replacement Surgery.
Brief Title: Pharmacokinetic (PK) Assessment of BIBR 1048 in Patients After Primary Elective Total Hip Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.30
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

ARMS (1):
- BIBR 1048 capsule (Experimental)
  Interventions: Drug: BIBR 1048 capsule

INTERVENTIONS:
Drug: BIBR 1048 capsule

SUMMARY:
To determine the PK profile of a single dose 150 mg BIBR 1048, oral capsule, administered 1-3 hours post surgery in hip replacement patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo a primary elective total hip replacement
* Male or female being 18 years or older (women of child bearing potential may not be included)
* Patients weighing at least 40 kg
* Written informed consent for participation

Exclusion Criteria:

* Bleeding disorders, e.g. history of intracranial, intraocular, gastrointestinal or pulmonary bleeding, known thrombocytopenia, history of haemorrhagic stroke
* Known renal disease
* Known liver disease, alcohol or drug misuse
* Known malignancy
* Treatment with another study drug in the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2002-04; Primary Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration (Cmax) | pre dose, 1, 2, 4, 6-8, 10-18 and 24 hours post dose
time to maximum plasma concentration (Tmax) | pre dose, 1, 2, 4, 6-8, 10-18 and 24 hours post dose
total clearance of drug from plasma | pre dose, 1, 2, 4, 6-8, 10-18 and 24 hours post dose
terminal elimination constant | pre dose, 1, 2, 4, 6-8, 10-18 and 24 hours post dose
time of last measureable BIBR 953 ZW plasma concentration (Tf) | pre dose, 1, 2, 4, 6-8, 10-18 and 24 hours post dose
area under the plasma concentration time curve until Tf (AUC0-Tf) | pre dose, 1, 2, 4, 6-8, 10-18 and 24 hours post dose
area under the plasma concentration time extrapolated to infinity (AUC0-infinity) | pre dose, 1, 2, 4, 6-8, 10-18 and 24 hours post dose

SECONDARY OUTCOMES:
Occurrence of adverse events | up to 24 hours after drug administration